CLINICAL TRIAL: NCT05834920
Title: Effects of Neurofeedback and Transcranial Pulse Stimulation on Attention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Maria Teresa Wijaya, Post-doctoral Fellow, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKUNFBTPS
Record Dates: First submitted 2023-03-17; First posted 2023-04-28 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Attention Difficulties
MeSH Terms: interventions — Transcranial Magnetic Stimulation; Neurofeedback

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neurofeedback (Active Comparator)
  Interventions: Device: Neurofeedback
- Transcranial pulse stimulation (Experimental)
  Interventions: Device: Transcranial pulse stimulation (TPS)
- Waitlist (No Intervention)

INTERVENTIONS:
Device: Transcranial pulse stimulation (TPS) — Participants will be treated with the TPS device NEUROLITH (Storz Medical AG). Treatments will be administered for up to 12 sessions within 4 weeks, each session consisting of 6000 TPS pulses of 0.2 mJ/mm².
  Arms: Transcranial pulse stimulation
Device: Neurofeedback — Participants will engage in a neurofeedback game designed to increase the ratio of theta/beta frequency bands in electroencephalography measurement. This intervention will be delivered for up to 12 sessions within 4 weeks.
  Arms: Neurofeedback

SUMMARY:
The present study aims to examine and compare the effectiveness of transcranial pulse stimulation and neurofeedback among adults who are weak in attention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years and above
* Right-handed
* Normal/corrected hearing and vision
* Having basic literacy skills
* Having sustained attention scores below the threshold

Exclusion Criteria:

* Having medical history related to brain
* Having mild cognitive impairment
* Showing symptoms of depression and anxiety
* Having intellectual disability based on IQ scores
* Having diagnoses of any psychiatric or cognitive disorders besides attention deficit hyperactivity disorder (ADHD) inattentive and combined types
* Having long-term history of smoking cigarettes
* Engaged in alcohol and/or substance abuse
* Having history of hemophilia or other blood clotting disorders or thrombosis
* Having corticosteroid treatment within the last six weeks before first intervention
* Having contraindications for MRI scanning

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Conners' Continuous Performance Test 3rd Edition | Baseline, week 4, week 8, week 12, week 16
  The Conners' Continuous Performance Test (CPT) measures inattentiveness, impulsivity, sustained attention, and vigilance. Participants are required to push the spacebar when any letter, except "X", appears. Performances are measured in raw scores and standardized T scores. T scores between 45-54 indicate average performance, higher or lower scores indicate atypical performance.
Change from baseline in gradCPT continuous performance test | Baseline, week 4, week 8, week 12, week 16
  The GradCPT is a continuous performance test to measure sustained attention. It has been shown to reliably indicate attentional fluctuation over time. Participants are required to respond to frequently presented city scene and inhibit responses to infrequently presented mountain scene. The sequence of visual stimuli is presented with gradual transitions to minimize involuntary attention capture by abrupt stimulus onset and offset. The main outcome of interest is reaction times variability, with higher variability indicating poorer sustained attention.

SECONDARY OUTCOMES:
Change from baseline in Stroop task | Baseline, week 4, week 8, week 12, week 16
  The Victoria version of the Stroop task is a validated means of measuring the ability to inhibit cognitive interference. Over three tasks of increasing difficulty level, participants are asked to identify colors as they appear on stimulus flash cards. These colors are randomly ordered either as dots, noncolor words, or noncorresponding color words. Performance is measured by reaction times and accuracy. Shorter reaction times and higher accuracy indicate better ability to inhibit cognitive interference.
Change from baseline in General Health Questionnaire | Baseline, week 4, week 8, week 12, week 16
  The General Health Questionnaire (GHQ) measures psychological well-being. It comprises 12 self-report questions, each assessing the severity of a mental problem over the past few weeks. Total scores range from 0 to 36 with a higher score indicating poorer psychological states.
Change from baseline in Goal Orientation Scale | Baseline, week 4, week 8, week 12, week 16
  The Goal Orientation Scale measures how individuals interpret and respond to achievement situations. It comprises three subscales. The present study uses only the learning goal orientation subscale which consists of 5 self-report items measuring the desire to develop the self by acquiring new skills, mastering new situations, and improving one's competence. Total scores range from 5 to 35 with higher scores indicating greater learning goal orientation.
Change from baseline in N-back task | Baseline, week 4, week 8, week 12, week 16
  The N-back task measures working memory function. Participants are presented a sequence of numbers ranging from 0 to 9 one-by-one. For each, they are required to decide whether the current stimulus is the same as the one presented two trials ago. Performance is measured by reaction times and accuracy. Shorter reaction times and higher accuracy indicate better working memory.
Change from baseline in Color Trails Test | Baseline, week 4, week 8, week 12, week 16
  The Color Trails Test (CTT) is used to assess attention shifting (i.e., the ability to alternate attention between two goals) and processing speed (i.e., the speed with which a cognitive operation is carried out). The test comprises two parts: CTT1 requires participants to connect a series of numbered circles that are randomly printed on a sheet of paper and CTT2 requires participants to connect numbered circles from 1 to 25 alternating between two colors (pink and yellow). Performance is measured by reaction times with faster reaction times indicating better flexibility and speed.
Change from baseline in Attentional Control Scale | Baseline, week 4, week 8, week 12, week 16
  The Attentional Control Scale is a self-report measure of attentional control. It consists of two subscales which measure selective attention and attention shifting respectively. Total scores range from 20 to 80 with higher scores indicating better attentional control.
Change from baseline in Rosenberg Self-esteem Scale | Baseline, week 4, week 8, week 12, week 16
  The Rosenberg Self-Esteem Scale is a 10-item self-report questionnaire which measures global self-esteem by measuring both positive and negative feeling about the self. Scores range from 10 to 40 with higher scores reflecting higher self-esteem.
Change from baseline in Social Connectedness Scale | Baseline, week 4, week 8, week 12, week 16
  The Social Connectedness Scale comprises 8 self-report items measuring three aspects of belongingness: connectedness, affiliation, and companionship. Total scores range from 8 to 48 with higher scores indicating higher sense of social connectedness.
Change from baseline in Hospital Anxiety and Depression Scale (HADS) | Baseline, week 4, week 8, week 12, week 16
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report questionnaire comprising two subscales which assess levels of anxiety and depression respectively. Total scores for each subscale range from 0 to 21 with higher scores indicating higher levels of anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- HKU InnoCentre of Clinical Neuropsychology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No